CLINICAL TRIAL: NCT04985721
Title: An Open Label, Signal Seeking, Translational, Phase II Trial of Pamiparib in Combination With Tislelizumab in Patients With Advanced Tumours With Homologous Recombination Repair Defects
Brief Title: A Trial of Pamiparib With Tislelizumab in Patients With Advanced Tumours With Homologous Recombination Repair Defects
Acronym: IMPARP-HRD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20/044
Record Dates: First submitted 2021-06-28; First posted 2021-08-02 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — pamiparib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pamiparib and Tiselizumab (Experimental)
  Interventions: Drug: Pamiparib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Pamiparib — 40 mg orally twice a day
Drug: Tislelizumab — 200 mg IV every 21 days

SUMMARY:
This study will describe the efficacy of pamiparib in combination with tislelizumab in patients with advanced tumours harbouring molecular profiles consistent with homologous recombination deficiency (HRD), agnostic of tumour origin. A tumour-agnostic approach has been adopted in this study due to the broad activity of PARP inhibitors across multiple tumour types. In addition, response to PARP inhibitors has been demonstrated in patients with genomic features associated with HRD, even in the absence of germline BRCA1 or BRCA2 mutations. These results suggest that the presence of HRD itself is the key predictive biomarker for PARP inhibitor efficacy. This paves the way for a precision-oncology, tumour-agnostic approach to patient selection for treatment, rather than the traditional tumour site-of-origin basis for which the current PARP inhibitor approvals exist. To investigate this, cohort A of this study includes patients with genomic features of HRD, but without a germline BRCA1 or BRCA2 mutation. Demonstration of clinical efficacy in this cohort will provide strong support to the tumour-agnostic, precision-oncology approach for patient selection for PARP inhibitor or PARP inhibitor combination treatment. This forms the primary objective of the study. The study will consist of two cohorts, broadly, cohort A - patients without a pathogenic BRCA1 or BRCA2 mutation but with other germline or somatic mutations in other HRD genes; cohort B- patients with a pathogenic BRCA1 or BRCA2

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Male or female ≥ 18 years of age
3. Patient has documentation of at least 1 of the following genomic features associated with HRD

   * Cohort A - any of:

     * A germline or somatic genetic alteration that is known or suspected to be deleterious in one of the following HR-related genes (ATM, CDK12, PALB2, ARID1A, ATRX, BLM, BARD1, BRIP1, CHEK1, CHEK2, FANCA, FANCF, FANCG, FANCI, FANCL, FANCM, MSH2, NBN, RAD50, RAD51C, RAD51D, WRN)
     * A somatic genetic alteration that is known or suspected to be deleterious in BRCA1 or BRCA2
     * A prevalent mutational signature 3 as determined by WGS (≥ 20% of total mutations attributed)
     * The presence of a positive HRD status using a NGS assay that includes assessment for genomic instability
     * Cohort A excludes high grade serous ovarian cancer, TNBC, and prostate cancer
   * Cohort B - a pathogenic germline BRCA1 or BRCA2 mutation Note: Genomic features associated with HRD must have been determined from a sample obtained ≤ 12 months before the date of registration into this study with the exception of germline genetic alterations which can have been determined from a sample obtained at any time.
4. Patient agrees to the collection and use of their fresh tumour biopsy sample during screening for WGS Note: A fresh tumour biopsy not required for patients who have had WGS performed within 12 months prior to registration to the study
5. Continues to meet all the inclusion criteria as per the TRIAGE Framework protocol
6. Measurable disease, as defined by RECIST 1.1 (see Appendix 2)
7. Adequate haematological and end-organ function, defined by the following laboratory results obtained within 7 days prior to registration, independent of blood or platelet transfusion within 2 weeks:

   * Haemoglobin ≥ 90 g/L
   * ANC ≥ 1.5x109/L
   * Platelet count ≥ 100 x109/L
   * ALT ≤ 3.0 x the ULN, irrespective of the presence or absence of liver metastases
   * AST ≤ 3.0 x the ULN, irrespective of the presence or absence of liver metastases
   * Serum bilirubin ≤ 1.5 x ULN (On fractionation ≤ 90% of total bilirubin should be unconjugated.

   Total bilirubin must be <4 x ULN for patients with Gilbert's Syndrome)
   * Serum creatinine ≤ 1.5x ULN or eGFR ≥ 30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (appendix 5)
   * INR ≤ 1.5x ULN (≤2.5x ULN if on anticoagulants)
8. Patient has the ability to take oral medications without medical history of malabsorption or other chronic gastrointestinal disease, or other conditions that may harm compliance and/or absorption of the study treatment
9. WOCBP must agree to use a highly effective method of birth control for the duration of the study and for 6 months after the last dose of study treatment (see Appendix 3), and have a negative serum pregnancy test within 7 days of study registration
10. Non-sterile males and their female partners must agree to use a highly effective method of birth control for the duration of the study and for 6 months after the last dose of study treatment. Non- sterile males must avoid sperm donation for the duration of the study and for at least 6 months after the last study drug
11. Female patient must agree not to breastfeed starting at screening and throughout the study period, and for 6 months after the final study drug administration
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing biopsies, treatment, and scheduled visits and examination including follow up

Exclusion Criteria:

1. One or more of the exclusion criteria as per the TRIAGE Framework protocol applies
2. Any previous treatment with a PARP inhibitor

   Note: Prior immune checkpoint blockade is permitted provided all the criteria below are met:
   * Patients must not have received the immune checkpoint blockade within 28 days of study registration
   * Patients must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy
   * All AEs while receiving prior immunotherapy must have completely resolved or resolved to grade

     1 prior to screening for this study. Patients with an endocrine AE due to immunotherapy are permitted provided they are stably maintained on appropriate replacement therapy and are asymptomatic
   * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not require maintenance doses of > 10 mg prednisolone or equivalent per day
3. Any unresolved toxicity (≥CTCAE grade 2) from previous anti-cancer therapy, with the exception of alopecia Note: Patients with irreversible toxicity that is not reasonably expected to be exacerbated by the study treatment (e.g. hearing loss, peripheral neuropathy) are eligible
4. Treatment with strong CYP3A inducers within 10 days (or ≤ 5 half-lives, whichever is shorter) prior to registration. Known need for treatment with strong CYP3A4 inducers during study treatment.
5. Symptomatic or current history of actively progressing CNS metastases. Patients with a history of treated CNS lesions are eligible, provided that all of the following criteria are met:

   * Measurable disease per RECIST 1.1 must be present outside the CNS
   * In patients who have received CNS-directed therapy, there is no clinical evidence of interim progression between completion of CNS-directed therapy and registration to the study (radiological re-assessment is not required)
   * The patient has not received radiotherapy within 14 days prior to registration Note: Anticonvulsant therapy at a stable dose is permitted

   Note: Patients with asymptomatic brain metastases in which CNS-directed therapy is not indicated are eligible
6. History of leptomeningeal disease
7. Mean QTc ≥ 470 ms calculated from triplicate ECGs using Fredericia's Correction
8. Active autoimmune disease or history of autoimmune disease that may relapse, with the following exceptions:

   * Controlled type 1 diabetes
   * Hypothyroidism managed with no treatment other than with hormone replacement therapy
   * Controlled celiac disease
   * Skin disease not requiring systemic treatment (e.g. vitiligo, psoriasis, alopecia)
   * Any other disease that is not expected to recur in the absence of external triggering factors
9. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication within 2 weeks prior to registration, with the following exceptions:

   * Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent)
   * Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption
   * Short course (≤ 7 days) of corticosteroid prescribed prophylactically or for the treatment of a non- autoimmune condition
10. Positive HIV test at screening
11. Patients with active HBV (chronic or acute; defined as having a positive HBsAg test at screening) or HCV Note: Patients with a past or resolved HBV infection (defined as the presence of HBcAb and absence of HBsAg) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA
12. Patients with severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including active tuberculosis and COVID-19
13. Patients with a history of interstitial lung disease, non-infectious pneumonitis or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung diseases, etc.
14. History of non-viral hepatitis or cirrhosis
15. Any of the following cardiovascular criteria:

    * Current evidence of cardiac ischemia.
    * Current symptomatic pulmonary embolism.
    * Acute myocardial infarction ≤ 6 months prior to study registration.
    * Heart failure of New York Heart Association Classification III or IV (See Appendix 6) ≤ 6 months prior to study registration.
    * Grade ≥ 2 ventricular arrhythmia ≤ 6 months prior to study registration.
    * History of cerebrovascular accident within 6 months before first dose of study drugs.
16. Has been administered a live vaccine within 4 weeks prior to registration
17. Known sensitivity to any component of pamiparib and/or tislelizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical benefit rate (CBR) in patients with advanced tumours harbouring molecular profiles consistent with homologous recombination defeciency (HRD), without a known pathogenic germline BRCA1 or BRCA2 mutation. | 12 weeks after commencement of treatment
  CBR, defined as the proportion of patients with either objective response (partial response (PR) + complete response (CR)) as best response, or stable disease (SD) at 12 weeks post registration, as determined by the Investigator by RECIST 1.1 in cohort A

SECONDARY OUTCOMES:
Efficacy of pamiparib in combination with tislelizumab in patients with advanced tumours harbouring molecular profiles consistent with HRD, and without a known pathogenic germline BRCA1 or BRCA2 mutation | At the end of the study, approximately 4 years after the first participant commences treatment
  Efficacy will be measured by:
  * overall response rate (ORR) - defined as the proportion of patients with an objective response (partial response + complete response) as best response (as determined by the Investigator by RECIST 1.1)
Efficacy of pamiparib in combination with tislelizumab in patients with advanced tumours harbouring molecular profiles consistent with HRD, and without a known pathogenic germline BRCA1 or BRCA2 mutation | At the end of the study, approximately 4 years after the first participant commences treatment
  Efficacy will be measured by:
  -progression free survival (PFS) - defined as the time from first dose of study medication to the first occurrence of disease progression, as determined by the Investigator according to RECIST 1.1, or death from any cause, whichever occurs first
Efficacy of pamiparib in combination with tislelizumab in patients with advanced tumours harbouring molecular profiles consistent with HRD, and without a known pathogenic germline BRCA1 or BRCA2 mutation | At the end of the study, approximately 4 years after the first participant commences treatment
  Efficacy will be measured by:
  -overall survival (OS) - defined as the time from first dose of study medication to death from any cause
Evaluation of CBR of pamiparib in combination with tislelizumab in patients with advanced tumours harbouring molecular profiles consistent with HRD (independent of germline BRCA1 or BRCA2 mutation status) | 12 weeks post commencement of treatment
  CBR, defined as the proportion of patients with either objective response (partial response (PR) + complete response (CR)) as best response, or stable disease (SD) at 12 weeks post registration, as determined by the Investigator by RECIST 1.1 in cohort A and B
Severity of Treatment -Emergent Events (Safety of pamiparib in combination with tiselizumab) | At the end of the study, approximately 4 years after the first participant commences treatment
  Severity of adverse events as determined by NCI CTCAE 5.0
Determination of HRD phenotype as a predictor of response | At the end of the study, approximately 4 years after the first participant commences treatment
  A tumour based whole genome HRD assay will provide a binary outcome as to whether HRD is "present" or "absent". Logistic regression models will be used to compare CBR between patients with tumours that have HRD "present" vs "absent".

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Luen, MBBS, Principal Investigator — Peter MacCallum Cancer Institute
Locations (3):
- Australia (3):
  - St Vincent's Hospital, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No